CLINICAL TRIAL: NCT03644433
Title: Impact of Single Layer Versus Double Layer Uterine Closure on the Cesarean Scar Healing
Brief Title: Impact of Uterine Closure Techniques on the Cesarean Scar Thickness After Repeated Cesarean Section
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Ragıp Atakan Al, Professor in obstetrics And gynecology, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: B.30.2.ATA.0.01.00/4
Record Dates: First submitted 2018-07-06; First posted 2018-08-23 (Actual); Last update posted 2018-08-24 (Actual); Status verified 2018-08

CONDITIONS: Cesarean Section, Repeated; Cesarean, Uterine Scar Thickness; Cesarean, Residual Myometrial Thickness; Cesarean Section Complications; Cesarean Section; Complications, Wound, Dehiscence
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Single layer (Placebo Comparator): Single layer closure
  Interventions: Procedure: Single layer closure
- Double layer with resection (Active Comparator): Double layer closure after resection uterine scar
  Interventions: Procedure: Double layer closure after resection uterine scar

INTERVENTIONS:
Procedure: Single layer closure — Uterine incision will be approximated with continuous unlocked suture avoiding the inclusion endometrium and without trimming incision edges.
  Arms: Single layer
Procedure: Double layer closure after resection uterine scar — Uterine incision will be trimmed and old scar tissue will be removed. Then first, endometrium will be approximated by continuous unlocked suture mimicking subcuticular suture avoiding the inclusion of endometrium and second, upper part of myometrium will be approximated by a continuous unlocked suture.
  Arms: Double layer with resection

SUMMARY:
We compares two techniques of uterine closure on myometrium thickness at the site of uterine scar of women who underwent repeated cesarean section. We will evaluate myometrial thickness by transvaginal ultrasound six months after cesarean.

ELIGIBILITY:
Inclusion Criteria:

* previous two or three cesarean
* gestational weeks >=36 weeks

Exclusion Criteria:

* risk of obstetric haemorrhage
* suspicion or diagnosis placenta previa or accrete syndrome
* chorioamnionitis
* uterine myoma in the anterior uterine segment
* hysterotomy other than lower segment uterine incision at previous cesarean

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Estimated)
Dates: Start 2018-08-23 (Actual); Primary Completion 2019-04-30 (Estimated); Study Completion 2019-04-30 (Estimated)

PRIMARY OUTCOMES:
residual myometrial thickness | 6 months after cesarean
  Myometrial thickness at the uterine scar by transvaginal ultrasound

SECONDARY OUTCOMES:
residual myometrial thickness | 6 weeks after cesarean
  Myometrial thickness at the uterine scar by transvaginal ultrasound
Healing ratio | 6 months after cesarean
  residual myometrial thickness * 100 /total myometrial thickness above uterine scar
Healing ratio | 6 weeks after cesarean
  residual myometrial thickness * 100 /total myometrial thickness above uterine scar
Existence of cesarean scar defect | 6 months after cesarean
  The presence or absence of a cesarean scar defect that was defined as any unechogenic area visualised by transvaginal ultrasound at the site of the cesarean scar with a depth of at least 1 mm.
Existence of cesarean scar defect | 6 weeks after cesarean
  The presence or absence of a cesarean scar defect that was defined as any unechogenic area visualised by transvaginal ultrasound at the site of the cesarean scar with a depth of at least 1 mm.
Operation time | 10 minute after cesarean completed
  skin-to-skin operation time
Change in hemoglobin | 48 hours after cesarean
  Difference in haemoglobin measured preoperatively and postoperatively 48 hours
Blood product transfusion | One week after cesarean
  unite number of transfused packed erythrocyte
Maternal infectious morbidity | six weeks after cesarean
  prevalence of postpartum endometritis, skin wound dehiscence and post operative fever.
Length of hospitalization | One month after cesarean
  Duration in days

CONTACTS AND LOCATIONS:
Locations (1):
- Atatürk Üniversitesi araştırma Hastanesi, Erzurum, Turkey (Türkiye)

REFERENCES:
- [Derived] Ozler MR, Al RA. A prospective comparative study of single-layer versus double-layer uterine closure techniques on cesarean scar formation. BMC Pregnancy Childbirth. 2025 Aug 20;25(1):868. doi: 10.1186/s12884-025-08010-3. PMID 40836292